CLINICAL TRIAL: NCT01870427
Title: NEWTON: A Single-center Open Label Study Evaluating Intravitreal Aflibercept Injection (IAI) for Previously Treated Macular Edema Associated With Central Retinal Vein Occlusions
Brief Title: NEWTON: Aflibercept Injection for Previously Treated Macular Edema Associated With Central Retinal Vein Occlusions
Acronym: NEWTON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern California Retina Vitreous Associates (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Rahul Khurana, M.D., Principal Investigator, Northern California Retina Vitreous Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCRVA-2013-Newton-4-01
Record Dates: First submitted 2013-05-25; First posted 2013-06-06 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Macular Edema With Central Retinal Vein Occlusions
Keywords: Macular Edema; Central Retinal Vein Occlusion; CRVO; Aflibercept; VEGF Trap-Eye; Eylea; Ranibizumab; Bevacizumab
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (2.0 mg) (Experimental): Intravitreal Aflibercept (2.0 mg)
  Interventions: Drug: Aflibercept (2.0 mg)

INTERVENTIONS:
Drug: Aflibercept (2.0 mg) — Intravitreal Aflibercept (2.0 mg)
  Other Names: Eylea; VEGF Trap-EYE

SUMMARY:
The purpose of the study is to determine the effect of Intravitreal Aflibercept Injection (IAI) on previously treated Central Retinal Vein Occlusions (CRVOs) with other Anti-VEGF agents.

DETAILED DESCRIPTION:
This prospective, open-label, single-center, nonrandomized, investigator-sponsored clinical study seeks to investigate the visual outcomes of a treat and extend dosing regimen of intravitreal aflibercept injection for macular edema following CRVO. All patients will receive IAI 2 mg at baseline and Week 4. If the pre-defined extension criteria are met at the 4-week visit, and at any follow up visit, the patient will receive a mandated treatment, and the next visit will be extended by two weeks. If the extension criteria are not met on a follow-up visit, the treatment interval will be continued to be reduced by 1 week. If criteria are still not met despite treatment at the reduced interval, treatment will be administered as usual and follow up interval will continue to be reduced by 1 week until the criteria are met or a 4-week interval is reached. Treatment of IAI is rendered at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above with documented history of center-involved macular edema secondary to CRVO.
* Patients must have received treatment for at least 6 months before baseline, with 3 initial loading doses, and evidence of recurrence of edema when extended beyond 4 weeks.
* Protocol refracted ETDRS BCVA of 20/25 to 20/320 (73-24 letters).
* Willing and able to comply with clinic visits and study-related procedures.
* Provide signed informed consent.

Exclusion Criteria:

* Prior panretinal or macular laser photocoagulation
* Previous use of intraocular corticosteroids or use of periocular corticosteroids within the 3 months prior to day 1
* Prior treatment with systemic anti-VEGF agents
* Presence of iris neovascularization
* Vitreous hemorrhage in the Study Eye
* Traction retinal detachment, or preretinal fibrosis involving the macula
* Diabetic macular edema or diabetic retinopathy, defined as eyes of diabetic patients with more than 1 microaneurysm outside the area of the vein occlusion.
* Infectious blepharitis, keratitis, scleritis, or conjunctivitis.
* Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or autoimmune-associated uveitis in either eye.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure equal or greater than 30mmHg despite treatment with anti-glaucoma medication)
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g. advanced glaucoma, age-related macular degeneration, etc)
* Any concurrent intraocular condition in the study eye (e.g. glaucoma) that, in the opinion of the investigator, could either require medical or surgical intervention during the 52 weeks study period to prevent or treat visual loss that might result from that condition.
* Pregnant or breast-feeding women
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus, contraceptive sponge, foam or jelly, or diaphragm) *Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Duration of Intravitreal Aflibercept on Treatment Interval | 52 Weeks
  Mean number of weeks between each injection where there is no macular edema

SECONDARY OUTCOMES:
Change in Visual Acuity | 52 Weeks
  Mean change in EDTRS BCVA
Retinal Thickness | 52 Weeks
  Mean change in Central Subfoveal Thickness by OCT
Adverse Events | 52 Weeks
  Incidence and severity of ocular and systemic AE's
Number of Treatments | 52 Weeks
  Mean number of Intravitreal Injections

CONTACTS AND LOCATIONS:
Overall Officials: Rahul N Khurana, MD, Principal Investigator — Northern California Retina Vitreous Associates
Locations (1):
- Northern California Retina Vitreous Associates, Mountain View, California, United States

REFERENCES:
- [Background] Brown DM, Heier JS, Clark WL, Boyer DS, Vitti R, Berliner AJ, Zeitz O, Sandbrink R, Zhu X, Haller JA. Intravitreal aflibercept injection for macular edema secondary to central retinal vein occlusion: 1-year results from the phase 3 COPERNICUS study. Am J Ophthalmol. 2013 Mar;155(3):429-437.e7. doi: 10.1016/j.ajo.2012.09.026. Epub 2012 Dec 4. PMID 23218699
- [Background] Boyer D, Heier J, Brown DM, Clark WL, Vitti R, Berliner AJ, Groetzbach G, Zeitz O, Sandbrink R, Zhu X, Beckmann K, Haller JA. Vascular endothelial growth factor Trap-Eye for macular edema secondary to central retinal vein occlusion: six-month results of the phase 3 COPERNICUS study. Ophthalmology. 2012 May;119(5):1024-32. doi: 10.1016/j.ophtha.2012.01.042. Epub 2012 Mar 21. PMID 22440275
- [Background] Heier JS, Campochiaro PA, Yau L, Li Z, Saroj N, Rubio RG, Lai P. Ranibizumab for macular edema due to retinal vein occlusions: long-term follow-up in the HORIZON trial. Ophthalmology. 2012 Apr;119(4):802-9. doi: 10.1016/j.ophtha.2011.12.005. Epub 2012 Feb 1. PMID 22301066
- [Background] Campochiaro PA, Brown DM, Awh CC, Lee SY, Gray S, Saroj N, Murahashi WY, Rubio RG. Sustained benefits from ranibizumab for macular edema following central retinal vein occlusion: twelve-month outcomes of a phase III study. Ophthalmology. 2011 Oct;118(10):2041-9. doi: 10.1016/j.ophtha.2011.02.038. Epub 2011 Jun 29. PMID 21715011
- [Derived] Khurana RN, Chang LK, Bansal AS, Palmer JD, Wu C, Wieland MR. Treat and extend regimen with aflibercept for chronic central retinal vein occlusions: 2 year results of the NEWTON study. Int J Retina Vitreous. 2019 Apr 15;5:10. doi: 10.1186/s40942-019-0159-x. eCollection 2019. PMID 31016030